CLINICAL TRIAL: NCT02333630
Title: Randomized Prospective Trial of a Mobile Health Application for Asthma Self-Management
Acronym: AsthmaCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Stukus (Other)
Responsible Party: Sponsor-Investigator, David Stukus, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB14-00678
Record Dates: First submitted 2014-12-17; First posted 2015-01-07 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AsthmaCare intervention (Experimental): Participants randomized to this arm will have the AsthmaCare app downloaded to their mobile device at time of study recruitment. They will have access to AsthmaCare indefinitely after enrollment.
  Interventions: Other: AsthmaCare mobile health application
- Control group (Active Comparator): Participants randomized to this arm will receive a link to a website containing asthma education videos and information. They will be able to access this link at their discretion.
  Interventions: Other: Asthma education

INTERVENTIONS:
Other: AsthmaCare mobile health application — Personalized, interactive mobile health application designed to send daily medication reminders and assist with self management
  Arms: AsthmaCare intervention
Other: Asthma education — A website with links to written asthma education and videos
  Arms: Control group

SUMMARY:
The investigators aim to study the clinical efficacy of a mobile health application, AsthmaCare, and it's impact on long term health outcomes for asthma. AsthmaCare is a novel application developed by members of the study team that was previously studied in a pilot study of 21 children/teenagers 9-16 years old. During the 30 day pilot study, there was universal usage and acceptance by all participants of this novel form of technology and asthma management. This current study aims to measure clinical outcomes for users of the app.

DETAILED DESCRIPTION:
AsthmaCare is a novel mobile health application that integrates personalized asthma reminders with self management feedback. Users input their prescribed daily controller medications and personal asthma triggers upon first loading the app. Reminder messages are pushed through the device at predetermined times to take controller medications. Once daily push notifications are sent to the user regarding tips to avoid preselected asthma triggers.

Users are asked to input their use of controller medications, which is entered into a medication log. Every interaction will unlock reward points as gaming theory is integrated into AsthmaCare to maintain user engagement.

If symptoms occur or if rescue medication use is logged into AsthmaCare, the user is automatically directed to an interactive asthma self-management plan, aka written asthma treatment plan. When users are in the yellow zone, they receive notifications every 4 hours regarding symptom update or rescue medication use. When users are in the red zone, these notifications occur every 1 hour. When users are in the green zone (baseline, no symptoms), they will receive motivational messages every 24 hours to maintain engagement with the app as well as remind them to continue to use controller medications.

In addition to medication reminders and an interactive self-management plan, AsthmaCare provides links to the nearest National Pollen Bureau counting station and allows for symptom/medication diaries to be emailed for sharing with providers or printing.

Mobile health applications, particularly for asthma, have not been studies in prospective clinical trials to demonstrate ongoing user engagement or efficacy. This study aims to determine whether users of an asthma mobile health application will have superior clinical outcomes compared with traditional asthma management.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of persistent asthma defined by treatment with at least one daily controller medication
* Fluent English speaking
* Subject must have access to an iOS or Android device in order to download and use the mobile health application
* At least one Emergency Department or Urgent Care visit due to asthma exacerbation in the 12 months prior to enrollment

Exclusion Criteria:

* No prescription/recommendation to use a daily controller medication
* Non-English speaking
* Lack of access to an iOS or Android device
* Current or prior use of AsthmaCare mobile health application at any time. Research assistant will assess by reviewing beforehand a complete list of people who have already downloaded the app

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Stukus, M.D., Principal Investigator — Nationwide Children's Hospital

REFERENCES:
- [Background] Martinez-Perez B, de la Torre-Diez I, Lopez-Coronado M. Mobile health applications for the most prevalent conditions by the World Health Organization: review and analysis. J Med Internet Res. 2013 Jun 14;15(6):e120. doi: 10.2196/jmir.2600. PMID 23770578
- [Background] Huckvale K, Car M, Morrison C, Car J. Apps for asthma self-management: a systematic assessment of content and tools. BMC Med. 2012 Nov 22;10:144. doi: 10.1186/1741-7015-10-144. PMID 23171675
- [Background] Free C, Phillips G, Galli L, Watson L, Felix L, Edwards P, Patel V, Haines A. The effectiveness of mobile-health technology-based health behaviour change or disease management interventions for health care consumers: a systematic review. PLoS Med. 2013;10(1):e1001362. doi: 10.1371/journal.pmed.1001362. Epub 2013 Jan 15. PMID 23349621
- [Background] Marcano Belisario JS, Huckvale K, Greenfield G, Car J, Gunn LH. Smartphone and tablet self management apps for asthma. Cochrane Database Syst Rev. 2013 Nov 27;2013(11):CD010013. doi: 10.1002/14651858.CD010013.pub2. PMID 24282112
- [Background] Chan AH, Reddel HK, Apter A, Eakin M, Riekert K, Foster JM. Adherence monitoring and e-health: how clinicians and researchers can use technology to promote inhaler adherence for asthma. J Allergy Clin Immunol Pract. 2013 Sep-Oct;1(5):446-54. doi: 10.1016/j.jaip.2013.06.015. Epub 2013 Aug 30. PMID 24565615
- [Derived] Stukus DR, Farooqui N, Strothman K, Ryan K, Zhao S, Stevens JH, Cohen DM. Real-world evaluation of a mobile health application in children with asthma. Ann Allergy Asthma Immunol. 2018 Apr;120(4):395-400.e1. doi: 10.1016/j.anai.2018.02.006. Epub 2018 Feb 13. PMID 29452259

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AsthmaCare Intervention | Control Group
Started | 100 | 100
Completed | 95 | 98
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AsthmaCare Intervention | Control Group | Total
Number analyzed (Participants) | 98 | 95 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.84 (5) | 6.24 (4.2) | 6.80 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 36 | 80
  Male | 54 | 59 | 113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 77 | 69 | 146
  White | 14 | 16 | 30
  More than one race | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 98 | 95 | 193
Insurance Provider [Count of Participants; unit: Participants]
  Medicaid | 86 | 93 | 179
  Commercial | 5 | 1 | 6
  Self pay | 7 | 1 | 8
Controller medications [Count of Participants; unit: Participants]
  Low dose ICS | 30 | 41 | 71
  Medium dose ICS | 28 | 20 | 48
  ICS and LABA | 10 | 7 | 17
  Montelukast | 1 | 1 | 2
  ICS and montelukast | 17 | 15 | 32
  ICS/LABA and montelukast | 12 | 11 | 23
Health Care Utilization for Asthma Exacerbations During 6 Months Prior to Enrollment [Mean (Standard Deviation); unit: visits]
  ED visits | 0.35 (0.56) | 0.29 (0.56) | 0.32 (0.55)
  Urgent Care visits | 0.3 (0.68) | 0.26 (0.57) | 0.28 (0.62)
  Hospitalizations | 0.17 (0.46) | 0.2 (0.5) | 0.19 (0.48)

OUTCOME MEASURES:

1. Primary Outcome: Number of Emergency Room Visits Secondary to Asthma Exacerbation
Description: Number of emergency room visits for asthma 6 months following study enrollment and randomization
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | AsthmaCare Intervention | Control Group
Number analyzed (Participants) | 98 | 95
visits | 0.31 (0.6) | 0.33 (0.74)

2. Secondary Outcome: Number of Asthma Exacerbations
Description: Number of prednisone courses prescribed for asthma exacerbations during 6 month study time frame
Time Frame: 6 months
Population: Data were not collected for this outcome measure
Groups:
- AsthmaCare: Participants randomized to AsthmaCare intervention
- Control: Participants randomized to control group
Arm/Group | AsthmaCare | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Hospitalizations
Description: Number of hospitalizations for asthma exacerbation during 6 month study duration
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | AsthmaCare Intervention | Control Group
Number analyzed (Participants) | 98 | 95
visits | 0.14 (0.38) | 0.1 (0.33)

4. Secondary Outcome: Frequency of Use of the Mobile Health Application
Description: Analytics from within the mobile application will be measured to determine the frequency and usage patterns of the mobile health application by users during the study period
Time Frame: 6 months
Population: Data were not collected for this measure
Groups:
- AsthmaCare; Control: Data were not collected for this measure
Arm/Group | AsthmaCare | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | AsthmaCare Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/95
Other Adverse Events (participants affected / at risk) | 0/98 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes